CLINICAL TRIAL: NCT01329523
Title: A Non-Randomized Controlled Cross-Sectional Study to Compare Genetic Variations of IGF-I and IGF-II in Patients With Moderate to Severe Dementia and Younger Family Members, in Relation to Age-Matched Unaffected Controls
Brief Title: A Study to Compare Genetic Variations of IGF-I and IGF-II
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AIHBG-1370-IGF
Record Dates: First submitted 2011-01-10; First posted 2011-04-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-01

CONDITIONS: Dementia
Keywords: Dementia; Insulin-like growth factor; IGF; APO E4; Genetics
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subjects with AD: Subjects with a diagnosis of dementia
- Family Members: Younger biological family members of the patients with dementia
- Control Group: Individuals without dementia matched in age to the patients with a dementia diagnosis

SUMMARY:
The purpose of this study is to determine if insulin-like growth factors (IGF) play a role in the development of dementia, specifically Alzheimer's disease (AD). The study will compare results from genetic testing between patients with AD and two other groups: younger biological family members of the AD patients and individuals without AD matched by age to the AD patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 50 and 81 years old who have a diagnosis of dementia
* Men and women who are at least 18 years old and are biologically related to the study subject with dementia
* Control subjects must not have a diagnosis of dementia and must be matched in age to the study subjects with dementia

Exclusion Criteria:

* Biological family members of the dementia patient who are either younger than 17 years of age or older than the patient with dementia
* Biological family members with a diagnosis of dementia
* Age-matched control subjects with a diagnosis of dementia

Ages: 50 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are three groups of participants for this research study: one group will consist of individuals diagnosed with dementia; another group will consist of younger biological family members of the patients with dementia; and the third group will consist of individuals without dementia who are matched in age to the patients with dementia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Genetic polymorphisms of insulin-like growth factors | Single clinic visit (day 1)
  This study consists of a single clinic visit. After subject has completed the informed consent process and meets eligibility criteria, a blood sample and a saliva sample will be collected. Genetic results from this one-time specimen collection will be evaluated and compared with results from participants in the other two study groups. Outcomes will be measured comparatively.

SECONDARY OUTCOMES:
Genetic testing of Apolipoprotein (APO) E4 | Single clinic visit (day 1)
  This study consists of a single clinic visit. After subject has completed the informed consent process and meets eligibility criteria, a blood sample and a saliva sample will be collected. Genetic results from this one-time specimen collection will be evaluated and compared with results from participants in the other two study groups. Outcomes will be measured comparatively.

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Chakunta, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Russo VC, Gluckman PD, Feldman EL, Werther GA. The insulin-like growth factor system and its pleiotropic functions in brain. Endocr Rev. 2005 Dec;26(7):916-43. doi: 10.1210/er.2004-0024. Epub 2005 Aug 30. PMID 16131630
- [Background] Freude S, Schilbach K, Schubert M. The role of IGF-1 receptor and insulin receptor signaling for the pathogenesis of Alzheimer's disease: from model organisms to human disease. Curr Alzheimer Res. 2009 Jun;6(3):213-23. doi: 10.2174/156720509788486527. PMID 19519303
- [Background] Lichtenwalner RJ, Forbes ME, Bennett SA, Lynch CD, Sonntag WE, Riddle DR. Intracerebroventricular infusion of insulin-like growth factor-I ameliorates the age-related decline in hippocampal neurogenesis. Neuroscience. 2001;107(4):603-13. doi: 10.1016/s0306-4522(01)00378-5. PMID 11720784
- [Background] Bingham EM, Hopkins D, Smith D, Pernet A, Hallett W, Reed L, Marsden PK, Amiel SA. The role of insulin in human brain glucose metabolism: an 18fluoro-deoxyglucose positron emission tomography study. Diabetes. 2002 Dec;51(12):3384-90. doi: 10.2337/diabetes.51.12.3384. PMID 12453890
- [Background] de la Monte SM, Wands JR. Alzheimer-associated neuronal thread protein mediated cell death is linked to impaired insulin signaling. J Alzheimers Dis. 2004 Jun;6(3):231-42. doi: 10.3233/jad-2004-6304. PMID 15201478